CLINICAL TRIAL: NCT02290028
Title: Sentus QP - Extended CRT Evaluation With Quadripolar Left Ventricular Leads
Acronym: QP ExCELs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: BIOTRONIK received FDA approval to transition the ongoing Sentus QP Study to a new EP PASSION real-world data methodology.
Sponsor: Biotronik SE & Co. KG (Industry)
Collaborators: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR016
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: CRT-D therapy; quadripolar left ventricular lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sentus QP left ventricular lead (Other): Subjects consented and implanted with a Sentus QP left ventricular lead.
  Interventions: Device: Sentus QP left ventricular lead

INTERVENTIONS:
Device: Sentus QP left ventricular lead — Implantation of quadripolar left ventricular lead in patients with CRT-D indication
  Other Names: Sentus OTW QP L; Sentus OTW QP S; Sentus OTW QP S-xx/49; Sentus OTW QP L-xx/49

SUMMARY:
The QP ExCELs study is designed to confirm safety and efficacy of the BIOTRONIK Sentus OTW QP left ventricular leads to satisfy FDA requirements for regulatory approval of the leads in the US. The Sentus OTW QP leads received FDA approval on May 4, 2017.

Long-term safety of the BIOTRONIK Sentus OTW QP left ventricular leads will be confirmed during the ongoing post approval phase (US sites only).

A protocol update was implemented on September 6, 2019 to transition the long-term follow up for the ongoing Sentus QP Study to a new EP PASSION real-world data methodology.

ELIGIBILITY:
Inclusion Criteria:

* Standard CRT-D indication according to clinical routine
* De novo implantation or upgrade from existing ICD or pacemaker implant utilizing a BIOTRONIK CRT-D system with IS4 LV port and Sentus QP LV lead
* Patient is able to understand the nature of the clinical investigation and provide written informed consent
* Patient is able and willing to complete all routine study visits at the investigational site through 5 years of follow-up
* Patient accepts Home Monitoring® concept
* Age ≥ 18 years

Exclusion Criteria:

* Chronic atrial fibrillation
* Contraindication to CRT-D therapy
* Currently implanted with an endocardial or epicardial left ventricular lead or had prior attempt to place a left ventricular lead
* Cardiac surgical procedure, such as coronary artery bypass graft or valve surgery that is planned to occur within 6 months after implant or ablation that is planned to occur within 90 days after implant (ablations planned to occur prior to or at implant are not exclusionary)
* Expected to receive a heart transplant or ventricular assist device within 6 months
* Life expectancy less than 12 months
* Participation in any other investigational cardiac clinical investigation during the course of the study
* Presence of another life-threatening, underlying illness separate from their cardiac disorder
* Pregnant or breast-feeding at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2226 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curnis, Prof., Study Chair — Spedali Civili - Universita di Brescia, Italy; Mattias Roser, Dr., Study Chair — Charité CBF Berlin, Germany
Locations (111):
- United States (67):
  - Fairhope, Alabama
  - Anchorage, Alaska
  - Chula Vista, California
  - Inglewood, California
  - Rancho Mirage, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Joliet, Illinois
  - Fort Wayne, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Bangor, Maine
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Fall River, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Ypsilanti, Michigan
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - Saint Charles, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Kalispell, Montana
  - Browns Mills, New Jersey
  - Englewood, New Jersey
  - Hackensack, New Jersey
  - Neptune City, New Jersey
  - Brooklyn, New York
  - Flushing, New York
  - New York, New York
  - The Bronx, New York
  - Valhalla, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Bryn Mawr, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wynnewood, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Amarillo, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Norfolk, Virginia
  - Milwaukee, Wisconsin
  - Cheyenne, Wyoming
- Australia (5):
  - Flinders Medical Center, Bedford Park
  - Lyell McEwing Hospital, Elizabeth Vale
  - The Northern Hospital, Epping
  - Royal Hobart Hospital, Hobart
  - Nambour General Hospital, Nambour
- Austria (3):
  - AKH Linz, Linz
  - AKH Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Denmark (2):
  - Gentofte Hospital, Hellerup
  - Odense Universitets Hospital, Odense
- Germany (21):
  - DHZ Berlin, Berlin
  - Maria Heimsuchung Caritas Klinik Pankow, Berlin
  - Virchow Klinikum, Berlin
  - Immanuel Klinikum Herzzentrum Bernau, Bernau
  - Städtisches Krankenhaus Bielefeld Mitte, Bielefeld
  - Augusta-Kranken-Anstalt Bochum, Bochum
  - Augusta Krankenhaus Düsseldorf, Düsseldorf
  - Heinrich Heine University Düsseldorf, Düsseldorf
  - Universitätsklinik Erlangen, Erlangen
  - Elisabeth Krankenhaus Essen, Essen
  - UHZ Freiburg, Freiburg im Breisgau
  - SRH Wald-Klinikum Gera gGmbH, Gera
  - Westpfalzklinikum, Kaiserslautern
  - Städtisches Klinikum St. Georg, Leipzig
  - UKSH Campus Lübeck, Lübeck
  - Marienhospital Lünen, Lünen
  - Elbekliniken Stade - Buxtehude, Stade
  - SBK Villingen Schwenningen, Villingen
  - SHG-Kliniken Völklingen, Völklingen
  - Universitätsklinikum Würzburg, Würzburg
  - HBK Zwickau, Zwickau
- Semmelweis University, Budapest, Hungary
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
- Italy (2):
  - Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Sant'Anna Como, Como
- Slovakia (2):
  - Nusch, Bratislava
  - Vusch East Slovak Cardiology Institute, Košice
- Spain (2):
  - Hospital Clinic Provincial de Barcelona, Barcelona
  - Hospital Ramón y Cajal Madrid, Madrid
- Switzerland (2):
  - Kantonspital Luzern, Lucerne
  - University Hospital Zürich, Zurich

RESULTS

PARTICIPANT FLOW:
Groups:
- Sentus QP Left Ventricular Lead: Participants consented and implanted with a Sentus QP left ventricular lead and CRT-D, plus participants that were consented but did not receive a Sentus QP lead or CRT-D.
Period: Overall Study
Arm/Group | Sentus QP Left Ventricular Lead
Started | 2226
Completed | 0
Not Completed | 2226
Not completed — Death | 217
Not completed — Sentus lead or required CRT-D was not implanted | 186
Not completed — No longer under care of study physician | 76
Not completed — Sentus lead or required CRT-D explanted | 55
Not completed — Withdrawal by Subject | 52
Not completed — Study site closure | 44
Not completed — Lost to Follow-up | 34
Not completed — Miscellaneous | 10
Not completed — Transition to EP PASSION | 1295
Not completed — Planned study completion at 12 months | 257

BASELINE CHARACTERISTICS:
Population: All participants consented with baseline data collection completed
Groups:
- Sentus QP Left Ventricular Lead: Participants consented and implanted with a Sentus QP left ventricular lead and CRT-D.
Arm/Group | Sentus QP Left Ventricular Lead
Number analyzed (Participants) | 2222
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Data collected and analyzed when available, not all subjects had data available for this measurement
  Years
    number analyzed (Participants) | 2221
    (all) | 68.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 683
  Male | 1539
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: Inches] — Population: Data collected and analyzed when available, not all subjects had data available for this measurement
  Inches
    number analyzed (Participants) | 2198
    (all) | 68.0 (4.0)
Weight [Mean (Standard Deviation); unit: Pounds] — Population: Data collected and analyzed when available, not all subjects had data available for this measurement
  Pounds
    number analyzed (Participants) | 2208
    (all) | 197.3 (50.0)

OUTCOME MEASURES:

1. Primary Outcome: Sentus QP Related Complication-free Rate Through 6 Months
Description: The purpose of primary endpoint 1 is to evaluate the Sentus QP related complication-free rate through 6 months post-implant. This is evaluated as a percentage of participants without a complication.
Time Frame: 6 months
Population: All participants in the Pre-Market cohort, defined as the study participants who were consented and implanted with a Sentus QP LV lead on or before January 29, 2016.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sentus QP Left Ventricular Lead
Number analyzed (Participants) | 279
percentage of participants | 97.1 [94.4 to 98.8]
Statistical Analysis 1: Comparison: Sentus QP Left Ventricular Lead; Primary endpoint 1 was evaluated by performing an exact, binomial test comparing the observed proportion (overall complication-free rate at 6 months) to the performance goal of 90.0%, with Type I error (alpha) of 0.025 and power of 80%. The lower, two-sided 95% confidence bound for the overall complication-free rate must be greater than 90.0%; Test type: Superiority; p < 0.0001, Exact, binomial

2. Primary Outcome: Percentage of Participants With Acceptable Pacing Threshold of Sentus QP Lead in Permanently Programmed Vector at 3 Months
Description: The purpose of primary endpoint 2 is to evaluate the LV lead pacing threshold for the permanently programmed pacing vector at 3 months post-implant.This was evaluated by performing an exact, binomial test comparing the percentage of participants with acceptable pacing thresholds to a performance goal of 88%. LV threshold values of less than or equal to 2.5 V at 0.4 ms in the permanently programmed vector are considered acceptable.
Time Frame: 3 months
Population: All participants in the Pre-Market cohort, defined as the study participants who were consented and implanted with a Sentus QP LV lead on or before January 29, 2016, and with completed threshold testing at 3 months post-implant or with available data from remote monitoring or next visits (as pre-specified in the protocol).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sentus QP Left Ventricular Lead
Number analyzed (Participants) | 286
percentage of participants | 93.4 [89.8 to 96.0]
Statistical Analysis 1: Comparison: Sentus QP Left Ventricular Lead; Primary endpoint 2 was evaluated by performing an exact, binomial test comparing an observed proportion (rate of acceptable LV pacing thresholds at the permanently programmed pacing vector at 3 months) to 88%, with Type I error (alpha) of 0.025 and power of 80%. The lower, two-sided 95% confidence bound for the percentage of subjects with an acceptable LV pacing threshold in the permanently programmed pacing vector must be greater than 88.0%; Test type: Superiority; p = 0.002, Exact, binomial

3. Primary Outcome: Sentus QP Related Complication-free Rate
Description: The purpose of primary endpoint 3 is to evaluate the Sentus QP related complication-free rate through study termination (post approval phase). This is evaluated as a percentage of participants without a complication.
Time Frame: Up to 4 years
Population: All participants in the Post-Market cohort, which included all participants who were enrolled with planned 5 year follow-up and were successfully implanted with a Sentus QP left ventricular lead.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sentus QP Left Ventricular Lead
Number analyzed (Participants) | 1727
percentage of participants | 98.03 [97.38 to 98.69]
Statistical Analysis 1: Comparison: Sentus QP Left Ventricular Lead; Primary endpoint 3 will be evaluated by performing an exact, binomial test comparing the observed proportion (overall complication-free rate at 5 years) to the performance goal of 92.5%, with Type I error (alpha) of 0.025 and power of 80%. The lower, two-sided 95% confidence bound for the overall complication-free rate must be greater than 92.5%; Test type: Superiority; On September 24, 2019, BIOTRONIK received FDA approval to transition the ongoing Sentus Post Approval Registry to a new EP PASSION real-world data methodology. As of study closure, the number of subjects with complete data required to perform the hypothesis test was not met. Therefore, this outcome measure was not analyzed

4. Secondary Outcome: Sentus QP Acceptable Pacing Threshold in Permanently Programmed Vector at 3 Months Per Lead Model
Description: The purpose of the secondary endpoint is to evaluate the LV lead pacing threshold for the permanently programmed pacing vector at 3 months post-implantation in the two different lead types, Sentus OTW QP L and Sentus OTW QP S. This was evaluated as the number of participants with an acceptable pacing threshold out of the total number of patients for each lead model. LV threshold values of less than or equal to 2.5 V at 0.4 ms in the permanently programmed vector is considered acceptable.
Time Frame: 3 months
Population: All participants in the Pre-Market cohort, defined as the study participants who were consented and implanted with a Sentus QP LV lead on or before January 29, 2016, and with completed threshold testing at 3 months post-implant.
Measure: Count of Participants; unit: Participants
Groups:
- Sentus QP L Model Left Ventricular Lead: Participants consented and implanted with a Sentus QP L model left ventricular lead and CRT-D.
- Sentus QP S Model Left Ventricular Lead: Participants consented and implanted with a Sentus QP S model left ventricular lead and CRT-D.
Arm/Group | Sentus QP L Model Left Ventricular Lead | Sentus QP S Model Left Ventricular Lead
Number analyzed (Participants) | 240 | 36
Participants | 226 | 32

5. Secondary Outcome: Sentus QP Acceptable Pacing Threshold in Novel Vectors at 3 Months
Description: The purpose of this secondary endpoint is to evaluate the number of participants with at least one acceptable LV lead pacing threshold in a novel pacing vector at 3 months post-implantation. This was evaluated as the number of participants with at least one acceptable LV pacing threshold in a novel pacing vector out of the total number of participants with completed novel pacing threshold testing. LV threshold values of less than or equal to 2.5 V at 0.4 ms in a novel pacing vector is considered acceptable.
Time Frame: 3 months
Population: All participants in the Pre-Market cohort, defined as the study participants who were consented and implanted with a Sentus QP LV lead on or before January 29, 2016, and with completed novel vector threshold testing at 3 months post-implant.
Measure: Count of Participants; unit: Participants
Arm/Group | Sentus QP Left Ventricular Lead
Number analyzed (Participants) | 273
Participants | 261

6. Secondary Outcome: Sentus QP Acceptable R-wave Sensed Amplitude at 3 Months Per Lead Model
Description: The purpose of this secondary endpoint is to evaluate acceptable LV lead sensing amplitude at 3 months post-implantation. This was evaluated as the number of participants with an acceptable LV sensing amplitude out of the total number of participants. R-wave sensed mean amplitude of greater than or equal to 2 mV is considered acceptable.
Time Frame: 3 months
Population: All participants in the Pre-Market cohort, defined as the study participants who were consented and implanted with a Sentus QP LV lead on or before January 29, 2016, and with completed sensing test at 3 months post-implant.
Measure: Count of Participants; unit: Participants
Arm/Group | Sentus QP L Model Left Ventricular Lead | Sentus QP S Model Left Ventricular Lead
Number analyzed (Participants) | 223 | 32
Participants | 223 | 32

7. Secondary Outcome: Sentus QP Acceptable Pacing Impedance at 3 Months Per Lead Model
Description: The purpose of this secondary endpoint is to evaluate the acceptable LV lead pacing impedance at 3 months post-implantation. This was evaluated as the number of participants with an acceptable LV pacing impedance out of the total participants. LV impedance values of greater than 200 Ohms and less than 2000 Ohms is considered acceptable.
Time Frame: 3 months
Population: All participants in the Pre-Market cohort, defined as the study participants who were consented and implanted with a Sentus QP LV lead on or before January 29, 2016, and with completed impedance testing at 3 months post-implant.
Measure: Count of Participants; unit: Participants
Arm/Group | Sentus QP L Model Left Ventricular Lead | Sentus QP S Model Left Ventricular Lead
Number analyzed (Participants) | 245 | 36
Participants | 245 | 36

8. Secondary Outcome: Sentus QP Time to Complication
Description: The purpose of this secondary is to evaluate the Sentus related complication-free rate through 6 months post-implant by the Kaplan-Meier method. The below table shows Kaplan-Meier estimates of the estimated freedom from Sentus related complications at 180 days.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sentus QP Left Ventricular Lead
Number analyzed (Participants) | 279
percentage of participants | 97.1 [95.14 to 99.13]

9. Secondary Outcome: Sentus QP Related Complication-free Rate Per Lead Model
Description: The purpose of secondary endpoint 7 is to evaluate the Sentus QP related complication-free rate through study termination (post approval phase). This is evaluated as percentage of participants without a complication per lead model.
Time Frame: Up to 4 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Sentus QP S Model Left Ventricular Lead: Participants consented and implanted with a Sentus QP S model left ventricular lead CRT-D.
Arm/Group | Sentus QP L Model Left Ventricular Lead | Sentus QP S Model Left Ventricular Lead
Number analyzed (Participants) | 1306 | 421
percentage of participants | 98.47 [97.80 to 99.13] | 96.67 [94.96 to 98.39]

10. Secondary Outcome: Individual Sentus QP Adverse Event Rates
Description: The purpose of secondary endpoint 8 is to evaluate the rate of individual types of adverse events related to the Sentus QP lead through study termination (post approval phase). This is evaluated as the percentage of participants with a specific adverse event out of the total participants.
Time Frame: Up to 4 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sentus QP Left Ventricular Lead
Number analyzed (Participants) | 1727
percentage of participants
  Dislodgements | 1.39 [0.08 to 1.94]
  Extracardiac Stimulation | 0.17 [0.04 to 0.51]
  Mechanical Lead Failure | 0.12 [0.01 to 0.42]
  Elevated Lead Impedance | 0.12 [0.01 to 0.42]
  Elevated LV Pacing Threshold | 0.06 [0.00 to 0.32]
  Electrical Lead Failure | 0.06 [0.00 to 0.32]
  Cardiac Perforation | 0.06 [0.00 to 0.32]

11. Secondary Outcome: Number of Participants Successfully Reprogrammed to Resolve Phrenic Nerve Stimulation or High Pacing Threshold
Description: The purpose of this secondary endpoint is to evaluate the number of participants in whom phrenic nerve stimulation or high LV pacing threshold was be successfully resolved by reprogramming of the LV pacing vector. This is evaluated as the number of participants with successful reprogramming out of all participants experiencing phrenic nerve stimulation or high LV pacing threshold. LV pacing threshold resulting in invasive intervention, or, in the absence of intervention, a lead threshold that has increased two fold from the chronic threshold value, and is unable to achieve a 2:1 safety margin at follow-up is considered a high LV pacing threshold.
Time Frame: 12 months
Population: All participants in the Pre-Market cohort, defined as the study participants who were consented and implanted with a Sentus QP LV lead on or before January 29, 2016, and whom experienced phrenic nerve stimulation or high LV pacing threshold.
Measure: Count of Participants; unit: Participants
Arm/Group | Sentus QP Left Ventricular Lead
Number analyzed (Participants) | 97
Participants | 73

ADVERSE EVENTS:
Time Frame: Though study exit or study termination, an average of 1.2 years, and up to 4 years
Description: According to the study protocol, sites were required to report all deaths and all adverse events that were considered related to the implant procedure, implanted pulse generator, or implanted leads. Adverse events determined to be not related to the implant procedure, implanted pulse generator, or implanted leads were not collected.
  Reported adverse events were defined as a serious or 'other' adverse event according to the clinicaltrials.gov definition.
Arm/Group | Sentus QP Left Ventricular Lead
All-Cause Mortality (participants affected / at risk) | 217/2226
Serious Adverse Events (participants affected / at risk) | 290/2226
Other Adverse Events (participants affected / at risk) | 711/2226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentus QP Left Ventricular Lead (N=2226)
Cardiac perforation associated with the RA lead (Cardiac disorders) | 1 (1)
Cardiac perforation associated with the RV lead (Cardiac disorders) | 3 (3)
Cardiac perforation associated with the LV lead (Cardiac disorders) | 1 (1)
Inability to place LV lead (Cardiac disorders) | 4 (4)
RA lead related lead dislodgement (Cardiac disorders) | 31 (31)
RV lead related lead dislodgement (Cardiac disorders) | 22 (23)
RV lead related elevated pacing threshold (Cardiac disorders) | 3 (3)
RV lead impedance out of range, high impedance (Cardiac disorders) | 3 (3)
RV lead related clinical failure (Cardiac disorders) | 3 (3)
RV lead related mechanical failure (Cardiac disorders) | 2 (2)
RV lead undersensing or loss of sensing (Cardiac disorders) | 1 (1)
Endocarditis associated with the RV lead (Cardiac disorders) | 1 (1)
LV lead related lead dislodgement (Cardiac disorders) | 59 (66)
LV lead related extracardiac stimulation (Cardiac disorders) | 11 (11)
LV lead related mechanical failure (Cardiac disorders) | 3 (3)
LV lead related high pacing threshold (Cardiac disorders) | 2 (2)
LV lead related elevated pacing threshold (Cardiac disorders) | 2 (2)
LV lead related clinical failure (Cardiac disorders) | 1 (1)
LV lead related loss of capture (Cardiac disorders) | 1 (1)
ICD device migration (Cardiac disorders) | 4 (4)
ICD device related inappropriate shock or ATP (Cardiac disorders) | 8 (8)
ICD device related electronic failure (Cardiac disorders) | 1 (1)
Twiddler's syndrome (General disorders) | 6 (6)
Implant procedure related infection (Infections and infestations) | 23 (24)
Secondary infection (Infections and infestations) | 10 (10)
Pocket infection (Infections and infestations) | 6 (6)
Cardiac perforation (Surgical and medical procedures) | 3 (4)
Arrhythmia associated with implant procedure (Surgical and medical procedures) | 7 (7)
Hematoma (Surgical and medical procedures) | 17 (17)
Loose set-screw (Surgical and medical procedures) | 1 (1)
Pneumothorax (Surgical and medical procedures) | 16 (16)
Pericarditis (Surgical and medical procedures) | 1 (1)
Pleural effusion (Surgical and medical procedures) | 4 (4)
Pericardial effusion (Surgical and medical procedures) | 2 (2)
Respiratory arrest (Surgical and medical procedures) | 1 (1)
Stroke (Surgical and medical procedures) | 1 (1)
Cardiogenic shock (Surgical and medical procedures) | 1 (1)
Respiratory distress (Surgical and medical procedures) | 3 (3)
Renal failure (Surgical and medical procedures) | 1 (1)
Wound healing disturbance (Surgical and medical procedures) | 3 (3)
Venous occlusion (Surgical and medical procedures) | 3 (3)
Discomfort/pain (Surgical and medical procedures) | 1 (1)
Post surgical bleeding (Surgical and medical procedures) | 5 (5)
Post procedure anemia (Surgical and medical procedures) | 2 (2)
Allergy to contrast agent (Surgical and medical procedures) | 1 (1)
Elevated WBD and labs post procedure (Surgical and medical procedures) | 1 (1)
Inflammation and swelling at surgical site (Surgical and medical procedures) | 1 (1)
RA lead elevated pacing threshold (Cardiac disorders) | 1 (1)
LV lead electrical lead failure (Cardiac disorders) | 1 (1)
LV lead impedance out of range, high (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentus QP Left Ventricular Lead (N=2226)
Inability to place LV lead (Cardiac disorders) | 101 (101)
RA lead related lead dislodgement (Cardiac disorders) | 7 (7)
RA lead related undersensing (Cardiac disorders) | 3 (3)
RV lead related clinical failure (Cardiac disorders) | 2 (2)
RV lead related extracardiac stimulation (Cardiac disorders) | 1 (1)
RV lead related high pacing threshold (Cardiac disorders) | 1 (1)
RV lead related oversensing (Cardiac disorders) | 1 (1)
LV lead related extracardiac stimulation (Cardiac disorders) | 258 (316)
LV lead related elevated pacing threshold (Cardiac disorders) | 132 (147)
LV lead related lead dislodgement (Cardiac disorders) | 27 (29)
LV lead related loss of capture (Cardiac disorders) | 24 (26)
LV lead impedance out of range, high impedance (Cardiac disorders) | 19 (20)
LV lead related high pacing threshold (Cardiac disorders) | 38 (40)
LV lead related clinical failure (Cardiac disorders) | 7 (7)
LV lead related oversensing (Cardiac disorders) | 4 (4)
LV lead related mechanical failure (Cardiac disorders) | 2 (2)
LV lead related electrical failure (Cardiac disorders) | 1 (1)
LV lead related loss of sensing (Cardiac disorders) | 1 (1)
ICD device migration (Cardiac disorders) | 1 (1)
ICD device related inappropriate shock or ATP (Cardiac disorders) | 6 (6)
ICD device related housing defect (Cardiac disorders) | 1 (1)
ICD device related high defibrillator (DFT) testing (Cardiac disorders) | 3 (3)
ICD device related pacemaker mediated tachycardia (PMT) (Cardiac disorders) | 2 (2)
Twiddler's syndrome (General disorders) | 3 (3)
Rachet syndrome (General disorders) | 1 (1)
Implant procedure related infection (Infections and infestations) | 8 (8)
Arrhythmia associated with implant procedure (Surgical and medical procedures) | 5 (5)
Hematoma (Surgical and medical procedures) | 12 (13)
Coronary sinus dissection (Surgical and medical procedures) | 9 (10)
Loose set-screw (Surgical and medical procedures) | 1 (1)
Pneumothorax (Surgical and medical procedures) | 3 (3)
Pericardial effusion (Surgical and medical procedures) | 4 (4)
Pleural effusion (Surgical and medical procedures) | 4 (4)
Bleeding at surgical site (Surgical and medical procedures) | 7 (7)
Allergy to surgery prep (Surgical and medical procedures) | 6 (6)
Unsuccessful defibrillator threshold (DFT) testing (Surgical and medical procedures) | 1 (1)
Wound healing disturbance (Surgical and medical procedures) | 5 (5)
Venous occlusion (Surgical and medical procedures) | 6 (6)
Discomfort/pain at surgical site (Surgical and medical procedures) | 14 (14)
RA lead elevated pacing threshold (Cardiac disorders) | 3 (4)
RA lead related extracardiac stimulation (Cardiac disorders) | 2 (3)
RA lead related thrombosis (Cardiac disorders) | 1 (1)
Pain in shoulder after system revision (Surgical and medical procedures) | 1 (1)
Hypotension after insertion procedure (Surgical and medical procedures) | 2 (2)
Bleeding caused by surgical prep (Surgical and medical procedures) | 1 (1)
Fever after insertion procedure (Surgical and medical procedures) | 1 (1)
Emesis after insertion procedure (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT02290028/Prot_SAP_000.pdf